CLINICAL TRIAL: NCT02163187
Title: Randomized Crossover Study of the Efficacy of Sacral Neuromodulation (SNM) With InterStimTM for Bowel Dysfunction Following Surgery for Rectal Cancers With Sphincter Preservation
Brief Title: Sacral Neuromodulation (SNM) With InterStimTM for Bowel Dysfunction Following Surgery for Rectal Cancers With Sphincter Preservation
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study permanently closed due to low accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14-100
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-01

CONDITIONS: Rectal Cancer; for Bowel Dysfunction Following Surgery for Rectal Cancers
Keywords: Neuromodulation (SNM); sphincter preservation; rectal polyp; InterStimTM; 14-100
MeSH Terms: conditions — Rectal Neoplasms | interventions — Leucine-tRNA Ligase; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- InterStimTM the device on (Experimental): The device will be set to stimulate for 4 weeks, then off for two weeks, and then the device will be on but will not stimulate for 4 weeks.
  Interventions: Device: Implantation of the InterStimTM; Behavioral: MSK BFI questionnaires; Behavioral: The Low Anterior Resection Score (LARS) questionnaires; Behavioral: The EuroQOL5D questionnaires; Behavioral: The Fecal incontinence Quality of Life Scale (FIQOL) questionnaires
- InterStimTM the device off (Experimental): The device will be on but will not stimulate for 4 weeks, then off for two weeks, and then the device will be set to stimulate for 4 weeks.
  Interventions: Device: Implantation of the InterStimTM; Behavioral: MSK BFI questionnaires; Behavioral: The Low Anterior Resection Score (LARS) questionnaires; Behavioral: The EuroQOL5D questionnaires; Behavioral: The Fecal incontinence Quality of Life Scale (FIQOL) questionnaires

INTERVENTIONS:
Device: Implantation of the InterStimTM
Behavioral: MSK BFI questionnaires
Behavioral: The Low Anterior Resection Score (LARS) questionnaires
Behavioral: The EuroQOL5D questionnaires
Behavioral: The Fecal incontinence Quality of Life Scale (FIQOL) questionnaires

SUMMARY:
The purpose of this study is to evaluate whether a medical device/implant (InterStimTM) will help patients to have more normal bowel movements. The InterStimTM device is a neuromodulating device. Neuromodulation is a way of changing the activity of the nervous system by using electrical stimulation. InterStimTM is FDA approved to help people who have a hard time controlling their bowl movements. This is called fecal incontinence.The device is placed near a nerve root in the lower back. It works in a manner similar to a pacemaker by releasing electrical stimulation that triggers the S3 nerve root. When being placed, it is initially tested to make sure it will work using a temporary wire and then, if successful, the device is permanently implanted.

DETAILED DESCRIPTION:
This is a single-blind randomized crossover study. After providing written informed consent, eligible patients will undergo an initial stimulation procedure with a temporary lead (Step 1 Wire Stimulation). The simulation is performed to determine efficacy of the device before a permanent implant is placed. This stimulation takes place over a period of 7-14 days (+/-3 days). Because this procedure is done in the OR, this window of time allows for optimization of the device and coordination of operating room schedules. This is the time period that has been used in prior trials. Typically bowel improvement has been seen relatively quickly, so the range should not affect our assessment of BFI.

After the Wire Implantation has occurred, patients will be evaluated over the next 7-14 days (+/- 3 days) and will complete the BFI questionnaire. If BFI improvement is < than or = to 4 points the wire will be removed in the operating room, the patient will be offered standard of care, and the patient will no longer be part of the study. Based on our prior data, we would like to give as many patients as possible the opportunity for enrollment and as a result we have chosen a 4 point BFI change as minimum criteria for response. Our group has seen that a change in the BFI around 5-6 is clinically significant, but we will lower this threshold slightly. If a patient's BFI improves by ≥ 4 points, the patient will proceed to the randomized phase (Step 2-Implantation) of the study.

Patients who proceed to Step 2- Implantation, they will return to the operating room for the implantation of the permanent device. While in the operating room they will be randomly assigned to either having the device stimulation on (Group A) or device stimulation off (Group B) for first 4 weeks (+/-3 days). Patients will return to clinic 2 weeks later to cross over to the other arm (Step 3-Crossover) and the device stimulation will be set to on or off. Patients will come back to clinic within 7 days (+/- 7 days) after Crossover for device check and optimization.

ELIGIBILITY:
Inclusion Criteria:

* History of rectal cancer or neoplastic polyp (i.e. intramucosal carcinoma, carcinoma in situ)
* BFI score must meet at least one of the below criteria:

  * Total BFI < 50
  * Dietary subscale < 11
  * Frequency subscale < 19
  * Urgency subscale < 12
* English speaking
* Patients ≥18 years old. age
* Sphincter-preserving surgery and ≥ 12 months after restoration of bowel continuity

Exclusion Criteria:

* Locally recurrent or metastatic disease
* Immune suppressive medication
* Seizure disorder
* Prior sacral/lower spinal surgery
* Congenital Spinal defect/Paraplegia
* Rectal prolapse
* IBD/Crohn's
* Pregnancy
* Active anal/rectal abscess
* Pacemaker or other electronic implanted device
* Immediate need for MRI
* At the time of the wire stimulation procedure, patients will be excluded if the surgeon is unable to place the temporary stimulating lead
* Inability to commit to local follow up for device management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06-10; Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Temple, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- InterStimTM the Device on, Then InterStimTM Device Off: The device will be set to stimulate for 4 weeks, then off for two weeks, and then the device will be on but will not stimulate for 4 weeks.
  Implantation of the InterStimTM
  MSK BFI questionnaires
  The Low Anterior Resection Score (LARS) questionnaires
  The EuroQOL5D questionnaires
  The Fecal incontinence Quality of Life Scale (FIQOL) questionnaires
- InterStimTM the Device Off, Then InterStimTM Device on: The device will be on but will not stimulate for 4 weeks, then off for two weeks, and then the device will be set to stimulate for 4 weeks.
  Implantation of the InterStimTM
  MSK BFI questionnaires
  The Low Anterior Resection Score (LARS) questionnaires
  The EuroQOL5D questionnaires
  The Fecal incontinence Quality of Life Scale (FIQOL) questionnaires
Period: Overall Study
Arm/Group | InterStimTM the Device on, Then InterStimTM Device Off | InterStimTM the Device Off, Then InterStimTM Device on
Started | 4 | 0
Treatment | 2 | 0
Completed | 2 | 0
Not Completed | 2 | 0
Not completed — Device removed | 1 | 0
Not completed — Progressive disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- InterStimTM the Device on, Then InterStim TM the Device Off: The device will be set to stimulate for 4 weeks, then off for two weeks, and then the device will be on but will not stimulate for 4 weeks.
- InterStimTM the Device Off, Then InterStim the Device on: The device will be on but will not stimulate for 4 weeks, then off for two weeks, and then the device will be set to stimulate for 4 weeks.
  No participants were accrued to this arm before the study was closed.
- Total: Total of all reporting groups
Arm/Group | InterStimTM the Device on, Then InterStim TM the Device Off | InterStimTM the Device Off, Then InterStim the Device on | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Continuous [Mean (Full Range); unit: years] | 53 [46 to 66] |  | 53 [46 to 66]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants were evaluable. 2 participants were non-evaluable.
  Participants
    Female | 3 |  | 3
    Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 4 |  | 4
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 4 |  | 4
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Bowel Function
Description: Bowel function will be assessed by using the MSK BFI. We have chosen the BFI because it is widely endorsed to assess the clinical problem that these patients have. The BFI is a 19 item instrument to which a patient responds using a 5-point Likert scale, ranging from Always to Never.
Time Frame: 3 years
Population: Study terminated early due to low accrual. Data were not collected.
Groups:
- InterStimTM the Device on: The device will be set to stimulate for 4 weeks, then off for two weeks, and then the device will be on but will not stimulate for 4 weeks.
  Implantation of the InterStimTM
  MSK BFI questionnaires
  The Low Anterior Resection Score (LARS) questionnaires
  The EuroQOL5D questionnaires
  The Fecal incontinence Quality of Life Scale (FIQOL) questionnaires
- InterStimTM the Device Off: The device will be on but will not stimulate for 4 weeks, then off for two weeks, and then the device will be set to stimulate for 4 weeks.
  Implantation of the InterStimTM
  MSK BFI questionnaires
  The Low Anterior Resection Score (LARS) questionnaires
  The EuroQOL5D questionnaires
  The Fecal incontinence Quality of Life Scale (FIQOL) questionnaires
Arm/Group | InterStimTM the Device on | InterStimTM the Device Off
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Quality of Life
Description: QOL and urinary continence will be assessed at the start of the study (Baseline), after initial stimulation (Step 1-Wire Stimulation), and at each point in the crossover trial (Step 2-Implantation and Step 3-Crossover). Graphical displays will be used to explore data distributions of all secondary outcome measures over time. We assume no period effect and will evaluate the treatment effect using the paired t-test (and a repeated measures ANOVA to include other covariates in the model) for each of our main outcome measures, EuroQOL5, FIQOL, LARS and Bladder function. We will test for period effect to confirm this.
Time Frame: 3 years
Population: Study terminated early due to low accrual. Data were not collected.
Arm/Group | InterStimTM the Device on | InterStimTM the Device Off
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: AE data not collected
Arm/Group | InterStimTM the Device on | InterStimTM the Device Off
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes